CLINICAL TRIAL: NCT05730101
Title: How to Help Students Overcome Academic Procrastination - Randomized-controlled Trial of Cognitive-behavioral Group and Imaginary Pills Treatment
Brief Title: How to Help Students Overcome Academic Procrastination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 024-22-01; ub23Heimgartner
Record Dates: First submitted 2023-01-27; First posted 2023-02-15 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Procrastination
Keywords: Academic procrastination; imaginary pill treatment; cognitive-behavioral treatment
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: three-arm randomized controlled trial with parallel group between-subject design
Masking Description: Blinding of participants and treatment providers is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No treatment waitlist group (No Intervention): Participants receive neither cognitive-behavioral nor imaginary pill treatment and are told that they are in the no treatment waitlist group. They are told that they can receive one of the treatments at the end of the study. The treatment they receive will be chosen based on study results.
- Cognitive-behavioral treatment group (CBT) (Active Comparator): Participants receive two individual and six group sessions with a therapist following the treatment manual "Prokrastination".
  Interventions: Other: Cognitive-behavioral treatment (CBT)
- Imaginary pill treatment group (IP) (Active Comparator): In accordance with the imaginary pill technique, participants are instructed to take an imaginary pill. This instruction consists of a procedure including five steps (i.e., 1) identifying the IP sensitive problem, 2) building trust/belief/reality of the IP, 3) constructing a personally meaningful IP, 4) taking the IP, 5) suggestions for self-administering the IP in real life and building adherence. The session is repeated with small modifications seven weeks later.
  Interventions: Other: Imaginary pill treatment (IP)

INTERVENTIONS:
Other: Cognitive-behavioral treatment (CBT) — In the first individual session (CBT1), together with the therapist, participants develop a behavioral and conditional model of their procrastination behavior. In the next 2 group sessions (CBT2 and CBT3), participants receive psychoeducation on procrastination. The focus is on learning the method of starting on time. In the third group session (CBT4), participants identify key procrastination-promoting thoughts and are supported to develop alternative thoughts; deepened in the second individual session (CBT5). In the next 2 group sessions (CBT 6 and CBT7), participants are informed about action planning with focus on learning to plan realistically. The last group session is a concluding session: Experiences with the methods learned and an outlook on further steps and goals are discussed. At the end of both individual sessions (CBT1 and CBT5), participants receive a link to an online survey to rate their treatment expectations (treatment expectation 1 and 2).
  Arms: Cognitive-behavioral treatment group (CBT)
Other: Imaginary pill treatment (IP) — In the first session (IP1), participants will be asked about the nature of their procrastination behavior and receive a procedure to take an imaginary pill following a rationale of 5 steps. In the second IP session (IP2), experiences with taking the IP are discussed and the procedure of taking the IP is adapted according to previous experiences and current needs. The rationale of the second session encompasses the same five steps with small modifications: 1) discussing IP sensitive problem and adapting it if necessary, 2) building trust/belief/reality of the IP, 3) discussing the personally meaningful IP and adapting it if necessary, 4) taking the IP, 5) adapting the procedure for self-administering the IP in real life on daily basis if necessary and building adherence. At the end of both sessions, participants receive a link to an online survey to rate their treatment expectations (treatment expectation 1 and 2).
  Arms: Imaginary pill treatment group (IP)

SUMMARY:
The purpose of this study is to evaluate two different treatment methods in a sample of procrastinating students of the University of Basel and the University of Applied Sciences and Arts Northwestern Switzerland. As first treatment, a cognitive-behavioral treatment has been chosen as these type of treatment already showed promising results in reducing students' procrastination behavior. The alternative to the more time-intensive cognitive-behavioral treatment is the application of imaginary pills to students suffering from procrastination.

This study evaluates the potential of the cognitive-behavioral and the imaginary pill treatment to reduce procrastination in a three-arm randomized controlled trial with parallel group between-subject design.

DETAILED DESCRIPTION:
Procrastination can be defined as "to voluntarily delay an intended course of action despite expecting to be worse off for the delay". Academic procrastination is limited to tasks and activities related to and/or relevant to learning and studying and manifests itself in consistently postponing studying for exams, submitting assignments late, and failing to register for classes in time. Despite the high prevalence of procrastination and the negative consequences on health and well-being, there is still no gold standard of treatment. The purpose of this study is to evaluate two different treatment methods in a sample of procrastinating students of the University of Basel and the University of Applied Sciences and Arts Northwestern Switzerland. As first treatment, a cognitive-behavioral treatment has been chosen as these type of treatment already showed promising results in reducing students' procrastination behavior. The alternative to the more time-intensive cognitive-behavioral treatment is the application of imaginary pills to students suffering from procrastination.

This study evaluates the potential of the cognitive-behavioral and the imaginary pill treatment to reduce procrastination in a three-arm randomized controlled trial with parallel group between-subject design.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Bachelor's and Master's students of the University of Basel and the University of Applied Sciences and Arts Northwestern Switzerland (FHNW)
* Age between 18 and 40
* Self-reported academic procrastination criterion is fulfilled (IPS value ≥ 29 points)
* Healthy by self-report statement (i.e., no known current physiological or psychological disorders, not taking medication, not in psychological/psychiatric treatment)
* Willing to participate in the study
* Sufficient German language skills to follow the instructions and participate in group sessions

Exclusion Criteria:

* Self-reported academic procrastination criteria not fulfilled: IPS < 29
* Any current psychological or physiological disease
* Current psychological or psychiatric treatment
* Current intake of psychotropic medication
* Insufficient German language skills to understand the instructions or discuss in group sessions
* Daily consumption of more than three alcoholic standard beverages (a standard alcoholic beverage is defined as either 3dl beer or 1dl wine or 2cl spirits)
* Regular drug consumption (THC, cocaine, heroin, etc.)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Change in German version of the Irrational Procrastination Scale (IPS) | At baseline (t0 = week 1), week 9 (t1), week 16 (t2), and week 42 (t4)
  Assessment of academic procrastination level: The IPS measures the degree of irrational delay causing procrastination. The German version of the IPS consists of nine questions, e.g. "I put things off so long that my well-being or efficiency unnecessarily suffers". Participants can respond on a 5-point scale ranging from 1="never" to 5="always/constantly".
Change in Academic Procrastination State Inventory (APSI) | At baseline (t0 = week 1), week 9 (t1), week 16 (t2), and week 42 (t4)
  Assessment of academic procrastination level: The APSI consists of 23 item, all referring to fluctuations in academic procrastination, behavior and thoughts and participants have to rate the frequency of engaging in the items in the previous week on a five point Likert scale ranging from 1="never" to 5="always".

SECONDARY OUTCOMES:
Change in Patient HealthQuestionnaire (PHQ-9) | At baseline (t0 = week 1), week 9 (t1), week 16 (t2), and week 42 (t4)
  Depressive symptoms are assessed with the Patient HealthQuestionnaire (PHQ-9). The PHQ-9 features nine items (e.g. "Little interest or enjoyment of your activities") to be rated on a four-point Likert scale (0="not at all" to 3="nearly every day").
Change in Generalized Anxiety Disorder Questionnaire-7 (GAD-7) | At baseline (t0 = week 1), week 9 (t1), week 16 (t2), and week 42 (t4)
  Anxiety is assessed with the Generalized Anxiety Disorder Questionnaire-7. It involves seven items assessing anxiety and excessive worry (e.g. "Feeling afraid as if something awful might happen") to be rated on a 4-point Likert scale (0="not at all" to 4="nearly every day").
Change in World Health Organization (WHO) Well-Being Index (WHO-5) | At baseline (t0 = week 1), week 9 (t1), week 16 (t2), and week 42 (t4)
  Subjective psychological well-being is assessed with the 5-item World Health Organization Well-Being Index (WHO-5). Items (e..g. "I have felt cheerful and in good spirits") are rated from 0="at no time" to 5="all the time".
Change in the German version of the Perceived Stress Scale (PSS-10) | At baseline (t0 = week 1), week 9 (t1), week 16 (t2), and week 42 (t4)
  Stress is assessed with the German version of the Perceived Stress Scale (PSS-10). 10 items assess the degree to which life has been experienced as unpredictable, uncontrollable and overwhelming (e.g. "In the last two weeks, how often have you felt nervous and stressed?"), rated on a 5-point Likert-type scale (0="never" to 4="very often").

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Heimgartner, lic. phil., Principal Investigator — University of Basel, Division of Clinical Psychologie and Psychotherapy, Faculty for Psychology
Locations (1):
- University of Basel, Division of Clinical Psychologie and Psychotherapy, Faculty for Psychology, Basel, Switzerland